CLINICAL TRIAL: NCT06023810
Title: The Effect of Watson's Human Care Theory-Based Motivational Interviewing on Treatment Adherence, Self-Efficacy, and Satisfaction in Individuals With Diabetic Foot Ulcers: A Randomized Controlled Trial
Brief Title: The Effect of Motivational Interviewing on Treatment Adherence, Self-Efficacy, and Satisfaction in Individuals With Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Collaborators: Sakarya University (Other)
Responsible Party: Principal Investigator, Nida Efetürk, Lecturer, Okan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IstanbulOkanU-N-EFETURK-001
Record Dates: First submitted 2023-08-10; First posted 2023-09-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Foot Ulcer, Diabetic
MeSH Terms: conditions — Diabetic Foot | interventions — Evaluation Studies as Topic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): Watson's human care theory-based motivational interviewing method
  Interventions: Behavioral: Watson's human care theory-based motivational interviewing method
- control (No Intervention)

INTERVENTIONS:
Behavioral: Watson's human care theory-based motivational interviewing method — The Motivational Interviewing Program based on Watson's Theory of Human Caring will be conducted over an 8-week period, with sessions taking place once a week. The initial session will have a duration of 60 minutes, while the subsequent weekly sessions will last for 30 minutes
  Other Names: Pre-post test
  Arms: experimental

SUMMARY:
The rise in diabetes incidence has led to a corresponding increase in diabetes-related complications. Diabetic foot ulcers, a severe consequence of diabetes, have substantial impacts on patients, the social environment, overall well-being, and nursing procedures. Given this context, there is a clear necessity for interventions that motivate patients to adopt beneficial health behaviors and educate them in effectively managing diabetes-related complications. This study seeks to investigate the impact of Watson's motivational interviewing method, which is grounded in the human care theory, on enhancing treatment adherence, self-efficacy, and satisfaction levels among individuals suffering from diabetic foot ulcers.

Hypotheses of The Research H0: There is no difference in self-efficacy for diabetic foot care, diabetic foot care behavior, treatment adherence, and satisfaction between individuals with diabetic foot ulcers who receive Watson's human care theory-based motivational interviewing and diabetic foot care education, and those who receive standard education.

H1: There is a difference in self-efficacy for diabetic foot care between individuals with diabetic foot ulcers who receive Watson's human care theory-based motivational interviewing and diabetic foot care education and those who receive standard education.

H2: There is a difference in diabetic foot care behavior between individuals with diabetic foot ulcers who receive Watson's human care theory-based motivational interviewing and diabetic foot care education and those who receive standard education.

H3: There is a difference in treatment adherence between individuals with diabetic foot ulcers who receive Watson's human care theory-based motivational interviewing and diabetic foot care education and those who receive standard education.

H4: There is a difference in satisfaction between individuals with diabetic foot ulcers who receive Watson's human care theory-based motivational interviewing and diabetic foot care education and those who receive standard education.

DETAILED DESCRIPTION:
According to the International Diabetes Federation (IDF) data, there are currently 425 million adults worldwide affected by diabetes, and it is projected to increase to 578 million by 2030 and 700 million by 2045. The increasing prevalence of diabetes has led to a rise in the frequency of complications arising from diabetes. The escalation in diabetes complications and their consequences is concerning. There is a need for interventions that encourage positive changes in health behaviors among patients and teach better management of diabetes-related complications.

Diabetic foot ulcer, a challenging complication of diabetes, has significant effects on physical, mental, social, and economic well-being, leading to reduced quality of life. It often necessitates prolonged hospitalizations, intensive treatment, and high medical costs. One of the nursing models frequently preferred today is the Human Care Theory, developed by Jean Watson between 1975 and 1979. The Human Care Theory is centered around providing quality care to patients and maintaining effective communication. Motivational Interviewing is a counseling approach developed by clinical psychologists William R. Miller and Stephen Rollnick.

The aim of the study is to investigate the impact of Watson's human care theory-based motivational interviewing method on treatment adherence, self-efficacy, and satisfaction in individuals with diabetic foot ulcers. In this study, a randomized controlled experimental-control group experimental design will be used. The population of the study consists of patients who applied to Kocaeli Derince Training and Research Hospital Internal Medicine outpatient clinics between June and October 2023, diagnosed with type 1 and type 2 diabetes mellitus, with first degree diabetic foot wound according to the Wagner classification. With the power analysis program G-Power 3.1.9.2, the sample size was calculated as 38 people (76) in each group.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with clear consciousness,
* No communication problems,
* Diagnosed with type 1 or type 2 diabetes,
* Grade 1 diabetic foot ulcer according to the Wagner classification,
* Receiving standard wound care,
* Residing in the Kocaeli province,
* No musculoskeletal or neurological disorders that could interfere with the study,
* Individuals willing to participate and who sign the informed consent form.

Exclusion Criteria:

- Patients who do not meet the inclusion criteria and those who decline to participate in the study will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Wagner's ulcer classification scale | at 1 week
  The Wagner classification divides ulcers based on the depth of the wound and the extent of gangrene. Grade 0, Skin intact but bony deformities lead to "foot at risk"; Grade 1, Superficial ulcer; Grade 2, Deeper, full thickness extension; Grade 3, Deep abscess formation or osteomyelitis; Grade 4, Partial Gangrene of forefoot; Grade 5; Extensive Gangrene.
Wagner's ulcer classification scale | at 8 weeks
  The Wagner classification divides ulcers based on the depth of the wound and the extent of gangrene. Grade 0, Skin intact but bony deformities lead to "foot at risk"; Grade 1, Superficial ulcer; Grade 2, Deeper, full thickness extension; Grade 3, Deep abscess formation or osteomyelitis; Grade 4, Partial Gangrene of forefoot; Grade 5; Extensive Gangrene.
Wagner's ulcer classification scale | at 12 weeks
  The Wagner classification divides ulcers based on the depth of the wound and the extent of gangrene. Grade 0, Skin intact but bony deformities lead to "foot at risk"; Grade 1, Superficial ulcer; Grade 2, Deeper, full thickness extension; Grade 3, Deep abscess formation or osteomyelitis; Grade 4, Partial Gangrene of forefoot; Grade 5; Extensive Gangrene.

SECONDARY OUTCOMES:
Diabetic Foot Care Self-Efficacy Scale | at 1 week
  It was developed to assess individuals' perception of their ability to perform diabetic foot care activities. The lowest score obtainable from the scale is 0, and the highest is 90. An increase in scale score indicates a higher level of individual self-efficacy.
Diabetic Foot Care Self-Efficacy Scale | at 8 weeks
  It was developed to assess individuals' perception of their ability to perform diabetic foot care activities. The lowest score obtainable from the scale is 0, and the highest is 90. An increase in scale score indicates a higher level of individual self-efficacy.
Diabetic Foot Care Self-Efficacy Scale | at 12 weeks
  It was developed to assess individuals' perception of their ability to perform diabetic foot care activities. The lowest score obtainable from the scale is 0, and the highest is 90. An increase in scale score indicates a higher level of individual self-efficacy.
Medication Adherence Report Scale | at 1 week
  The scale consists of 5 items rated on a 5-point Likert scale. Scores obtained from the items are summed to calculate the total test score. An increase in the total score obtained from the scale indicates agreement, while a decrease indicates disagreement
Medication Adherence Report Scale | at 8 weeks
  The scale consists of 5 items rated on a 5-point Likert scale. Scores obtained from the items are summed to calculate the total test score. An increase in the total score obtained from the scale indicates agreement, while a decrease indicates disagreement
Medication Adherence Report Scale | at 12 weeks
  The scale consists of 5 items rated on a 5-point Likert scale. Scores obtained from the items are summed to calculate the total test score. An increase in the total score obtained from the scale indicates agreement, while a decrease indicates disagreement
Watson Patient Satisfaction Assessment Form According to Healing Processes | at 8 weeks
  The form consists of a total of six questions. The first five questions are scored on a scale of 1 to 7, with responses ranging from 'never' (1) to 'always' (7).

CONTACTS AND LOCATIONS:
Locations (1):
- Derince Training and Research Hospital, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No